CLINICAL TRIAL: NCT00937040
Title: A Placebo Controlled Double-Blind, Parallel Group, Individualizing Dosing Study Optimizing Treatment of Adults With Attention Deficit Hyperactivity Disorder to an Effective Response With OROS Methylphenidate
Brief Title: Adult Study / OROS Methylphenidate Hydrochloride (HCL) (OROS MPH) in Adults With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR015058; CONCERTA-ATT-3014 (Other: Ortho-McNeil Janssen Scientific Affairs, LLC)
Record Dates: First submitted 2009-06-29; First posted 2009-07-10 (Estimated); Results first posted 2011-08-05 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Osmotic Release Oral System (OROS®) Extended Release Methylphenidate HCl; CONCERTA® (OROS MPH)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 001 (Experimental): OROS MPH Optimal Patient Dose (18 mg-72 mg) once daily by mouth for 6 weeks
  Interventions: Drug: OROS MPH; Drug: OROS MPH Tablets
- 002 (Placebo Comparator): Placebo Optimal Patient Dose (placebo to match 18 mg - 72 mg) once daily by mouth for 6 weeks
  Interventions: Drug: Placebo; Drug: Placebo Tablets

INTERVENTIONS:
Drug: OROS MPH — Optimal Patient Dose (18 mg-72 mg) once daily for 6 weeks
  Arms: 001
Drug: Placebo — Optimal Patient Dose (placebo to match 18 mg - 72 mg) once daily for 6 weeks
  Arms: 002
Drug: OROS MPH Tablets — Optimal Patient Dose (18 mg-72 mg) once daily by mouth for 6 weeks
  Arms: 001
Drug: Placebo Tablets — Optimal Patient Dose (placebo to match 18 mg - 72 mg) once daily by mouth for 6 weeks
  Arms: 002

SUMMARY:
The purpose of this study is to compare the ADHD symptom response of adults with ADHD treated with OROS MPH to those treated with placebo.

DETAILED DESCRIPTION:
The hypothesis is that Osmotic Release Oral System (OROS) Extended Release Methylphenidate HCL (OROS MPH) is safe and effective in improving Attention Deficit Hyperactivity Disorder (ADHD) symptoms in adults with ADHD when compared to placebo as demonstrated using specific study measures. This is a double-blind (neither participant nor investigator knows the name of the assigned study drug), randomized (study drug assigned by chance), placebo-controlled study to evaluate the efficacy and safety of OROS MPH using the optimal dose for each adult patient in the study with ADHD. The primary efficacy variable in this study is the change from baseline to final evaluation using the Adult ADHD Investigator Symptom Rating Scale (AISRS) to measure patient ADHD symptoms. Participants will also be assessed for adverse events throughout the study. Patients will initiate treatment with oral OROS MPH 18 mg or matching placebo at baseline and continue morning dosing with increases every week until an optimal dose is achieved, up to the maximum of 72 mg/day of OROS MPH or matching placebo. Eligible patients will remain in the study for a maximum of 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* ADHD diagnosis (any type: Combined, Predominantly Inattentive, or Predominantly Hyperactive-Impulsive)
* Patients with an Adult ADHD Investigator Symptom Rating Scale (AISRS) score greater than 24 at screening/baseline
* Ability to read and understand English

Exclusion Criteria:

* Any significant history of cardiovascular disease or cardiovascular disease detectable via ECG
* History of diagnosis of substance or alcohol dependence or admission/hospitalization for rehabilitation for dependence
* Current neurologic or psychiatric diagnosis that would make patient inappropriate for participation
* Anxiety assessments of moderate or severe
* Depression assessments of moderate or severe
* History or current suicidal thoughts or attempts
* Known allergies, hypersensitivity, or intolerance to OROS MPH

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2009-07; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ortho-McNeil Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Ortho-McNeil Janssen Scientific Affairs, LLC

REFERENCES:
- [Derived] Goodman DW, Starr HL, Ma YW, Rostain AL, Ascher S, Armstrong RB. Randomized, 6-Week, Placebo-Controlled Study of Treatment for Adult Attention-Deficit/Hyperactivity Disorder: Individualized Dosing of Osmotic-Release Oral System (OROS) Methylphenidate With a Goal of Symptom Remission. J Clin Psychiatry. 2017 Jan;78(1):105-114. doi: 10.4088/JCP.15m10348. PMID 27487193

RESULTS

PARTICIPANT FLOW:
Groups:
- PLACEBO: Once daily (morning) tablet(s) taken orally of 18, 36 , 54, or 72 mg of placebo
- OROS MPH: Once daily (morning) tablet(s) taken orally of 18, 36 , 54, or 72 mg of Osmotic Release Oral System (OROS) Extended Release Methylphenidate HCl (MPH) - CONCERTA
Period: Overall Study
Arm/Group | PLACEBO | OROS MPH
Started | 179 | 178
Completed | 138 | 141
Not Completed | 41 | 37
Not completed — Adverse Event | 5 | 8
Not completed — Lost to Follow-up | 12 | 12
Not completed — Protocol Violation | 3 | 0
Not completed — Withdrawal by Subject | 13 | 7
Not completed — NONCOMPLIANCE WITH STUDY DRUG | 3 | 2
Not completed — POST ENROLL EXCLUSIONARY LAB(S)/ECG FIND | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PLACEBO | OROS MPH | Total
Number analyzed (Participants) | 179 | 178 | 357
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 3 | 6
  Between 18 and 65 years | 175 | 173 | 348
  >=65 years | 1 | 2 | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 34.6 (11.53) | 36.8 (11.87) | 35.7 (11.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 86 | 165
  Male | 100 | 92 | 192
Region of Enrollment [Number; unit: participants]
  USA | 179 | 178 | 357

OUTCOME MEASURES:

1. Primary Outcome: Adult Attention Deficit Hyperactivity Disorder (ADHD) Investigator Symptom Rating Score (AISRS) Over Time Using the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) Fourth Edition for Diagnosis
Description: The Adult ADHD Investigator Symptom Rating Score (AISRS) assesses 18 core ADHD symptoms corresponding to the DSM-IV diagnostic symptoms for adult subjects based on the investigator's rating for each of the symptoms using a four point scale (0=None, 1=Mild, 2=Moderate, and 3=Severe). If a single item is missing the score is imputed and if more than one item is missing, the total score is treated as missing. The AISRS total score is derived by summing the score assigned to each of the 18 symptoms (low=0, high=54, a higher score signifies a greater severity of symptoms).
Time Frame: Baseline, endpoint (42 days or early discontinuation)
Population: Intent-to-Treat (ITT) analysis set was defined as all randomized subjects who have received at least one dose of the study medication and have any post-baseline efficacy data (not including ASRS).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PLACEBO | OROS MPH
Number analyzed (Participants) | 172 | 169
units on a scale
  Baseline | 37.0 (7.51) | 37.8 (6.94)
  Endpoint | 25.2 (13.47) | 20.7 (12.76)
  Change from baseline at endpoint | -11.7 (13.30) | -17.1 (12.44)
Statistical Analysis 1: Comparison: PLACEBO vs OROS MPH; Gate-Keeper-Sequence#01. The primary efficacy was tested at the 0.05 level of significance. To control the overall Type I error at 0.05, the secondary efficacy endpoints were tested in a fixed sequence if the preceding null hypothesis was rejected. No further hypotheses could be tested when the preceding null hypothesis was not rejected. All nominal p-values were presented even though the formal testing procedure stopped at the primary endpoint. No unqualified statements can be made; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was determined by using an ANCOVA model with factors treatment and pooled study center, and covariate baseline AISRS total score. Change from baseline to endpoint uses the latest non-missing score after baseline for each subject; P-value for Change from baseline at endpoint. Each outcome involved with gate-keeping will be numbered with a Gate-Keeper-Sequence-Number from 01-16

2. Secondary Outcome: Reaction Time Domain of the Stroop Test (Cognitive and Executive Function)
Description: Stroop Test is a computerized measure of inhibition/disinhibition, executive function, reaction time, and information processing. The 1st part generates basic "reaction time" to colors. The 2nd part generates "complex reaction time score" to matching color names and font color. The 3rd part establishes a "Stroop reaction time" and an error score to unmatched color names/fonts. Reaction Time Domain Score = (Stroop Complex Reaction Time Correct + Stroop Reaction Time Correct)/2. Lower scores indicate better functioning (i.e. reaction time).
Time Frame: Baseline, 4 hour timepoint for extended days or last non-missing value for non-extended days on day 42 or early discontinuation (endpoint)
Population: Intent-to-Treat (ITT) analysis set. Only non-missing values are shown at each category (timepoint). Change from baseline to endpoint requires a non-missing value at both baseline and endpoint.
Measure: Mean (Standard Deviation); unit: milliseconds (msec)
Arm/Group | PLACEBO | OROS MPH
Number analyzed (Participants) | 172 | 169
milliseconds (msec)
  Baseline (N=140,132) | 708.0 (134.36) | 700.3 (141.09)
  Endpoint (N=108,114) | 653.2 (108.68) | 645.2 (116.56)
  Change from baseline at endpoint (N=103,101) | -39.8 (118.16) | -51.2 (123.45)
Statistical Analysis 1: Comparison: PLACEBO vs OROS MPH; Gate-Keeper-Sequence-Number#02; Test type: Superiority or Other; p = 0.206, ANCOVA — P-value was determined by using an ANCOVA model with factors treatment and pooled study center, and covariate baseline score. Endpoint for extended day sites is the 4 hour timepoint and for other sites is the last non-missing value after baseline; P-value for Change from baseline at endpoint

3. Secondary Outcome: Vigilance Domain (Complex Attention) of the Stroop Test/Shifting Attention Test (SAT)/Continuous Performance Test (CPT) (Cognitive and Executive Function)
Description: The Stroop Test is a computerized measure of inhibition/disinhibition, executive function, reaction time, and information processing. The Shifting Attention Test (SAT) a computerized measure of the ability to shift from one instruction set to another quickly and accurately. The Continuous Performance Test (CPT) is a computerized measure of vigilance or sustained attention/attention over time. Vigilance Domain (Complex Attention) Score = Stroop Commission Errors + SAT Errors + CPT Commission Errors + CPT Omission Errors. Lower scores indicate better functioning (i.e. sustained attention).
Time Frame: Baseline, endpoint (42 days or early discontinuation)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: errors
Arm/Group | PLACEBO | OROS MPH
Number analyzed (Participants) | 172 | 169
errors
  Baseline (N=140,132) | 28.2 (39.43) | 35.7 (47.15)
  Endpoint (N=108,114) | 27.2 (43.97) | 23.9 (37.04)
  Change from baseline at endpoint (N=103,101) | -0.2 (47.98) | -10.4 (45.82)
Statistical Analysis 1: Comparison: PLACEBO vs OROS MPH; Gate-Keeper-Sequence-Number#03; Test type: Superiority or Other; p = 0.348, ANCOVA — [p-value comment as in outcome 2, analysis 1]; P-value for Change from baseline at endpoint

4. Secondary Outcome: Cognitive Flexibility Domain of the Stroop/SAT Tests (Cognitive and Executive Function)
Description: The Stroop Test is a computerized measure of inhibition/disinhibition, executive function, reaction time, and information processing. The SAT is a computerized measure of the ability to shift from one instruction set to another quickly and accurately. The scores generated by the SAT are: correct matches, errors, and response time. The testing score is a measure of cognitive flexibility. Cognitive Flexibility Domain Score = SAT Correct Responses - SAT Errors - Stroop Commission Errors. Higher scores indicate better accuracy.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: correct responses
Arm/Group | PLACEBO | OROS MPH
Number analyzed (Participants) | 172 | 169
correct responses
  Baseline (N=140,132) | 34.0 (21.54) | 31.5 (21.57)
  Endpoint (N=108,114) | 45.9 (17.40) | 46.6 (17.67)
  Change from baseline at endpoint (N=103,101) | 11.3 (18.86) | 13.9 (20.34)
Statistical Analysis 1: Comparison: PLACEBO vs OROS MPH; Gate-Keeper-Sequence-Number#04; Test type: Superiority or Other; p = 0.324, ANCOVA — [p-value comment as in outcome 2, analysis 1]; P-value for Change from baseline at endpoint

5. Secondary Outcome: Processing Speed Domain of the Symbol Digit Modalities Test (SDTM) (Cognitive and Executive Function)
Description: The Symbol Digit Modalities Test (SDMT) is a computerized variant of the Wechsler Digit Symbol Substitution Test (DSST), but the position of symbols and digits is reversed. Scoring is the number of correct responses generated in 2 minutes. Processing Speed Domain = SDMT correct responses - SDMT errors. Higher scores indicate better functioning (i.e. information processing).
Time Frame: Baseline, endpoint (42 days or early discontinuation)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: acccurate responses per minute
Arm/Group | PLACEBO | OROS MPH
Number analyzed (Participants) | 172 | 169
acccurate responses per minute
  Baseline (N=140,132) | 53.9 (12.65) | 52.8 (13.17)
  Endpoint (N=109,114) | 59.7 (13.23) | 58.8 (25.68)
  Change from baseline at endpoint (N=104,101) | 5.9 (9.14) | 4.9 (23.88)
Statistical Analysis 1: Comparison: PLACEBO vs OROS MPH; Gate-Keeper-Sequence-Number#05; Test type: Superiority or Other; p = 0.631, ANCOVA — [p-value comment as in outcome 2, analysis 1]; P-value for Change from baseline at endpoint

6. Secondary Outcome: Global Executive Composite (GEC) Score of the Brief Rating Inventory of Executive Function for Adults (BRIEF-A)
Description: The BRIEF-A is a self-reported measure (low=61, high=225, lower scores indicate higher executive functioning) capturing views of the subject's own functioning in the everyday environment. The BRIEF-A contains 75 scored items (1=never, 2=sometimes, 3=often) in 9 non-overlapping clinical scales (Inhibit, Shift, Emotional Control, Self-Monitor, Initiate, Working Memory, Plan/Organize, Task Monitor, and Organization of Materials). The Behavioral Regulation Index (BRI), Metacognition Index (MI), and GEC are then derived.
Time Frame: Baseline, endpoint (42 days or early discontinuation)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PLACEBO | OROS MPH
Number analyzed (Participants) | 172 | 169
units on a scale
  Baseline (N=168,166) | 153.3 (23.22) | 153.7 (19.73)
  Endpoint (N=157,155) | 137.9 (32.19) | 128.4 (28.98)
  Change from baseline at endpoint (N=153,153) | -14.5 (29.18) | -25.8 (26.97)
Statistical Analysis 1: Comparison: PLACEBO vs OROS MPH; Gate-Keeper-Sequence-Number#06; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was determined by using an ANCOVA model with factors treatment and pooled study center, and covariate baseline score; P-value for Change from baseline at endpoint

7. Secondary Outcome: Performance and Daily Functioning Scale of the Adult ADHD Impact Module (AIM-A)
Description: The AIM-A is a subject-reported measure (low=0, high=100, a higher score is more favorable) to assess the overall impact and role that ADHD may have in the conduct of tasks that are expected of adults. The AIM-A is comprised of four global quality of life items, five economic impact items, and five multi-item scales that describe important concepts. Items include: Living with ADHD; General Well-Being; Work, Home and School Performance and Daily Functioning; Relationships; and Communication; and Impact of Symptoms (emotional, degree of daily interference).
Time Frame: Baseline, endpoint (42 days or early discontinuation)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PLACEBO | OROS MPH
Number analyzed (Participants) | 172 | 169
units on a scale
  Baseline (N=168,166) | 36.0 (18.34) | 31.9 (17.45)
  Endpoint (N=157,155) | 48.5 (26.11) | 59.4 (24.14)
  Change from baseline at endpoint (N=153,153) | 12.7 (24.00) | 27.5 (26.44)
Statistical Analysis 1: Comparison: PLACEBO vs OROS MPH; Gate-Keeper-Sequence-Number#07; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 6, analysis 1]; P-value for Change from baseline at endpoint

8. Secondary Outcome: Subject's Rating of Endicott Work Productivity Scale (EWPS)
Description: The EWPS provides a measure of the subject's report of their overall productivity (low=0, high=100, a higher score indicates worsening work productivity and efficiency). There are 25 items (questions 15-39) on the scale that describe types of behaviors/ subjective feelings that are highly likely to reduce work productivity/efficiency. These 25 items are rated on a 5-point scale (0=never, 1=rarely, 2=sometimes, 3=often, to 4=almost always) indicating how often the behavior, feeling or attitude has been manifested in the past week. The total score is the sum of the 25 items.
Time Frame: Baseline, endpoint (42 days or early discontinuation)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PLACEBO | OROS MPH
Number analyzed (Participants) | 172 | 169
units on a scale
  Baseline (N=129,141) | 44.7 (19.68) | 46.2 (17.07)
  Endpoint (N=126,124) | 33.3 (21.70) | 27.6 (18.53)
  Change from baseline at endpoint (N=104,115) | -9.7 (20.58) | -18.0 (18.54)
Statistical Analysis 1: Comparison: PLACEBO vs OROS MPH; Gate-Keeper-Sequence-Number#08; Test type: Superiority or Other; p = 0.008, ANCOVA — [p-value comment as in outcome 6, analysis 1]; P-value for Change from baseline at endpoint

9. Secondary Outcome: Subject's Rating of Dyadic Satisfaction Subscale (DSS)
Description: The Dyadic Adjustment Scale (DAS) assesses the relationship satisfaction or adjustment of partners in committed couple relationships. The 32-question DAS includes 4 empirically validated subscales that measure: dyadic satisfaction, dyadic consensus, dyadic cohesion and affectional expression. The response format varies across the entire scale and includes 5-, 6-, and 7-point Likert-scale questions and two yes/no items. The 10-question subset of the DAS, the Dyadic Satisfaction Subscale, was used in this study (low=0, high=50, higher score means better relationship satisfaction).
Time Frame: Baseline, endpoint (42 days or early discontinuation)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PLACEBO | OROS MPH
Number analyzed (Participants) | 172 | 169
units on a scale
  Baseline (N=65,80) | 32.3 (6.92) | 31.4 (6.62)
  Endpoint (N=66,68) | 32.5 (7.57) | 33.3 (6.68)
  Change from baseline at endpoint (N=46,52) | 0.0 (4.88) | 1.4 (4.66)
Statistical Analysis 1: Comparison: PLACEBO vs OROS MPH; Gate-Keeper-Sequence-Number#09; Test type: Superiority or Other; p = 0.372, ANCOVA — [p-value comment as in outcome 6, analysis 1]; P-value for Change from baseline at endpoint

10. Secondary Outcome: Subject's Rating of Satisfaction With Treatment Questionnaire - Overall, How Satisfied or Dissatisfied Are You With the Medication You Are Taking for ADHD?
Description: The satisfaction with treatment questionnaire (low=0, high=20, a lower score indicates lower satisfaction with treatment) requires subjects to answer 4 questions related to how much their ADHD symptoms have changed since starting the medication, how much benefit they received from the medication, the extent, if any, the advantages outweighed the disadvantages, and overall satisfaction with the medication. The responses for this question vary with range of satisfaction (e.g. extremely satisfied, very satisfied, satisfied, neutral, dissatisfied, very dissatisfied, or extremely dissatisfied).
Time Frame: Endpoint (42 days or early discontinuation)
Population: Intent-to-Treat (ITT) analysis set for non-missing response to this question
Measure: Number; unit: Participants
Arm/Group | PLACEBO | OROS MPH
Number analyzed (Participants) | 157 | 155
Participants
  Extremely Dissatisfied | 39 | 14
  Very Dissatisfied | 18 | 17
  Dissatisfied | 24 | 7
  Neither Dissatisfied or Satisfied | 38 | 36
  Satisfied | 16 | 40
  Very Satisfied | 15 | 28
  Extremely Satisfied | 7 | 13
Statistical Analysis 1: Comparison: PLACEBO vs OROS MPH; Gate-Keeper-Sequence-Number#10; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — P-value was determined by using the Cochran-Mantel-Haenszel (CMH) row mean scores controlling for center; P-value for Change from baseline at endpoint

11. Secondary Outcome: Responder Rate Using AISRS
Description: AISRS responder rate is defined as the percentage of subjects with AISRS < 18 at endpoint.
Time Frame: Endpoint (42 days or early discontinuation)
Population: Intent-to-Treat (ITT) analysis set
Measure: Number; unit: Percent of participants
Arm/Group | PLACEBO | OROS MPH
Number analyzed (Participants) | 172 | 169
Percent of participants
  Responder | 30.8 | 45.0
  Non-responder | 69.2 | 55.0
Statistical Analysis 1: Comparison: PLACEBO vs OROS MPH; Gate-Keeper-Sequence-Number#11; Test type: Superiority or Other; p = 0.008, Cochran-Mantel-Haenszel — P-value was determined using CMH general association controlling for pooled center; P-value for Change from baseline at endpoint

12. Secondary Outcome: Clinical Global Impression - Severity of Illness Subscale (CGI-S)
Description: The Clinical Global Impression - Severity of Illness (CGI-S) is a clinician-rated subscale (low=0, high=7, higher score indicates increasing illness). The clinician rates the severity of the ADHD symptoms in relation to the clinician's total experience with ADHD subjects using a 7-point scale (1=normal, not at all ill, 2= borderline ill, 3= mildly ill, 4=moderately ill, 5= markedly ill, 6= severely ill, 7= among the most extremely ill subjects) in response to the question "Considering your total clinical experience with this particular population, how ill is the subject at this time?".
Time Frame: Baseline, endpoint (42 days or early discontinuation)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PLACEBO | OROS MPH
Number analyzed (Participants) | 172 | 169
units on a scale
  Baseline | 4.6 (0.69) | 4.7 (0.75)
  Endpoint (N=160,158) | 3.5 (1.28) | 3.0 (1.37)
  Change from baseline at endpoint (N=160,158) | -1.1 (1.33) | -1.7 (1.46)
Statistical Analysis 1: Comparison: PLACEBO vs OROS MPH; Gate-Keeper-Sequence-Number#12; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 6, analysis 1]; P-value for Change from baseline at endpoint

13. Secondary Outcome: Significant Other's (a Spouse, Significant Other or Other Adult in the Household, Described in This Study as the Designated Observer) Rating of Adult ADHD Rating Scale IV
Description: The ADHD Rating Scale-IV (Significant Other) is an 18-item list of core ADHD symptoms corresponding to the DSM-IV diagnostic symptoms. Each item is rated on a four point Likert type scale (0 = never or rarely, 1 = sometimes, 2 = often, and 3 = very often). The subject's designated observer will complete this scale, with baseline assessment based on the subject's usual functioning when not on medication. The total score is derived by summing the score assigned to each of the 18 symptoms (low=0, high=54, a higher score signifies a greater severity of symptoms).
Time Frame: Baseline, endpoint (42 days or early discontinuation)
Population: Intent-to-Treat (ITT) analysis set and non-missing values at each timepoint. Only non-missing values are shown at each category (timepoint). Change from baseline to endpoint requires a non-missing value at both baseline and endpoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PLACEBO | OROS MPH
Number analyzed (Participants) | 59 | 54
units on a scale
  Baseline (N=51,40) | 29.9 (12.19) | 29.2 (12.00)
  Endpoint (N=40,35) | 27.3 (12.01) | 21.7 (13.75)
  Change from baseline at endpoint (N=35,28) | -1.7 (9.77) | -8.3 (10.90)
Statistical Analysis 1: Comparison: PLACEBO vs OROS MPH; Gate-Keeper-Sequence-Number#13; Test type: Superiority or Other; p = 0.003, ANCOVA — [p-value comment as in outcome 6, analysis 1]; P-value for Change from baseline at endpoint

14. Secondary Outcome: Designated Observer's (DO) Global Executive Composite (GEC) Score of the Brief Rating Inventory of Executive Function for Adults (BRIEF-A)
Description: The BRIEF-A, as completed by the DO, is a measure (low=61, high=225, lower scores indicate higher executive functioning) capturing views of an adult informant familiar with the subject's functioning. The BRIEF-A contains 75 scored items (1=never, 2=sometimes, 3=often) in nine non-overlapping clinical scales (Inhibit, Shift, Emotional Control, Self-Monitor, Initiate, Working Memory, Plan/Organize, Task Monitor, and Organization of Materials). The Behavioral Regulation Index (BRI), Metacognition Index (MI), and Global Executive Composite (GEC) are then derived.
Time Frame: Baseline, endpoint (42 days or early discontinuation)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PLACEBO | OROS MPH
Number analyzed (Participants) | 80 | 76
units on a scale
  Baseline (N=66,58) | 139.3 (27.08) | 144.1 (24.77)
  Endpoint (N=55,52) | 133.3 (26.54) | 127.3 (27.18)
  Change from baseline at endpoint (N=44,39) | -10.3 (19.79) | -20.1 (26.25)
Statistical Analysis 1: Comparison: PLACEBO vs OROS MPH; Gate-Keeper-Sequence-Number#14; Test type: Superiority or Other; p = 0.016, ANCOVA — [p-value comment as in outcome 6, analysis 1]; P-value for Change from baseline at endpoint

15. Secondary Outcome: Designated Observer's (DO) Rating of Dyadic Satisfaction Subscale
Description: The Dyadic Adjustment Scale (DAS) completed by DOs who were spouses or significant others assesses the relationship satisfaction or adjustment of partners in committed couple relationships. The 32-question DAS includes 4 empirically validated subscales that measure: dyadic satisfaction, dyadic consensus, dyadic cohesion and affectional expression. Possible responses include 5-, 6-, and 7-point Likert-scale questions and two yes/no items. The 10-question DAS subset, the Dyadic Satisfaction Subscale, was used in this study (low=0, high=50, higher score means better relationship satisfaction).
Time Frame: Baseline, endpoint (42 days or early discontinuation)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PLACEBO | OROS MPH
Number analyzed (Participants) | 80 | 76
units on a scale
  Baseline (N=44,43) | 36.2 (6.75) | 35.8 (8.29)
  Endpoint (N=43,38) | 37.5 (6.08) | 37.2 (8.38)
  Change from baseline at endpoint (N=31,31) | 0.6 (4.32) | 1.5 (4.16)
Statistical Analysis 1: Comparison: PLACEBO vs OROS MPH; Gate-Keeper-Sequence-Number#15; Test type: Superiority or Other; p = 0.092, ANCOVA — [p-value comment as in outcome 6, analysis 1]; P-value for Change from baseline at endpoint

16. Secondary Outcome: Designated Observer's (DO) Rating of Satisfaction With Treatment Questionnaire - Overall, How Satisfied or Dissatisfied Are You With the Medication for ADHD Your Partner is Taking?
Description: The satisfaction with treatment questionnaire (low=0, high=20, a lower score indicates lower satisfaction with treatment) requires the subject's DO to answer 4 questions related to how much the subject's ADHD symptoms have changed since starting the medication, how much benefit was received from the medication, the extent, if any, the advantages outweighed the disadvantages, and overall satisfaction with the medication. Responses vary from extremely satisfied, very satisfied, satisfied, neutral, mildly dissatisfied, dissatisfied, very dissatisfied, or extremely dissatisfied.
Time Frame: Endpoint (42 days or early discontinuation)
Population: Intent-to-Treat (ITT) analysis set for non-missing response to this question
Measure: Number; unit: Participants
Arm/Group | PLACEBO | OROS MPH
Number analyzed (Participants) | 80 | 76
Participants
  Extremely Dissatisfied | 5 | 2
  Very Dissatisfied | 4 | 2
  Dissatisfied | 8 | 6
  Neither Dissatisfied or Satisfied | 19 | 9
  Satisfied | 5 | 10
  Very Satisfied | 6 | 3
  Extremely Satisfied | 0 | 0
  Missing/Unknown | 33 | 44
Statistical Analysis 1: Comparison: PLACEBO vs OROS MPH; Gate-Keeper-Sequence-Number#16; Test type: Superiority or Other; p = 0.284, Cochran-Mantel-Haenszel — P-value was determined by using the Cochran-Mantel-Haenszel (CMH) row mean scores controlling for center. Missing/unknown responses are not included in the p-value; P-value for Change from baseline at endpoint

17. Secondary Outcome: Adult ADHD Self-Report Scale (ASRS) Over Time
Description: The Adult ADHD Self-Report Scale (ASRS) assesses 18 core ADHD symptoms corresponding to the DSM-IV diagnostic symptoms for adult subjects based on the subject's own rating for each of the symptoms using a four point scale (0=None, 1=Mild, 2=Moderate, and 3=Severe). If a single item is missing the score is imputed and if more than one item is missing, the total score is treated as missing. The ASRS total score is derived by summing the score assigned to each of the 18 symptoms (low=0, high=54, a higher score signifies a greater severity of symptoms).
Time Frame: Baseline, endpoint (42 days or early discontinuation)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PLACEBO | OROS MPH
Number analyzed (Participants) | 172 | 169
units on a scale
  Baseline (N=167, 166) | 49.8 (10.11) | 51.6 (9.73)
  Endpoint (N=171,167) | 37.5 (16.33) | 32.6 (16.04)
  Change from baseline at endpoint (N=166, 165) | -12.1 (15.86) | -19.4 (15.86)
Statistical Analysis 1: Comparison: PLACEBO vs OROS MPH; P-value for Change from baseline at endpoint; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 6, analysis 1]

18. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI) Total Score
Description: The PSQI discriminates between good and poor sleepers. The self-administered scale contains 15 multiple-choice items concerning frequency of sleep disturbances and subjective sleep quality and 4 write-in items that inquire about typical bedtime, wake-up time, sleep latency, and sleep duration over the past month. The PSQI generates 7 scores corresponding to the different sleep domains. Each component score ranges from 0 to 3. Total sleep index is calculated by adding up the 7 component scores (low=0, high=21, the lower the score, the better in sleep quality).
Time Frame: Baseline, endpoint (42 days or early discontinuation)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PLACEBO | OROS MPH
Number analyzed (Participants) | 172 | 169
units on a scale
  Baseline (N=167, 166) | 8.8 (3.47) | 9.1 (3.17)
  Endpoint (N=157, 155) | 8.5 (3.25) | 8.4 (3.14)
  Change from baseline at endpoint (N=152, 153) | -0.4 (3.00) | -0.8 (2.96)
Statistical Analysis 1: Comparison: PLACEBO vs OROS MPH; P-value for Change from baseline at endpoint; Test type: Superiority or Other; p = 0.319, ANCOVA — [p-value comment as in outcome 6, analysis 1]

19. Secondary Outcome: Epworth Sleepiness Scale (ESS)
Description: The Epworth Sleepiness Scale (ESS) is an 8-item self-rated questionnaire designed to assess the overall level of daytime sleepiness. Each item describes normal daily situations (i.e., watching TV, lying down in the afternoon, sitting inactive in a public place) and subjects rate the likelihood of dozing off or falling asleep in each situation. Responses use a 4-point rating scale (0=would never doze, 1=slight chance of dozing, 2=moderate chance of dozing, 3=high chance of dozing). Item scores are summed to produce a total score (range of 0-24) with lower score suggesting more alertness.
Time Frame: Baseline, endpoint (42 days or early discontinuation)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PLACEBO | OROS MPH
Number analyzed (Participants) | 172 | 169
units on a scale
  Baseline (N=167,166) | 9.1 (5.01) | 9.5 (4.81)
  Endpoint (N=157,155) | 8.0 (5.20) | 7.0 (4.86)
  Change from baseline at endpoint (N=152,153) | -1.0 (4.56) | -2.5 (4.13)
Statistical Analysis 1: Comparison: PLACEBO vs OROS MPH; P-value for Change from baseline at endpoint; Test type: Superiority or Other; p = 0.007, ANCOVA — [p-value comment as in outcome 6, analysis 1]

ADVERSE EVENTS:
Arm/Group | PLACEBO | OROS MPH
Serious Adverse Events (participants affected / at risk) | 1/175 | 0/174
Other Adverse Events (participants affected / at risk) | 49/175 | 100/174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PLACEBO (N=175) | OROS MPH (N=174)
Suicidal Ideation (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PLACEBO (N=175) | OROS MPH (N=174)
Headache (Nervous system disorders) | 20 | 33
Nausea (Gastrointestinal disorders) | 8 | 9
Dry Mouth (Gastrointestinal disorders) | 3 | 27
Upper Respiratory Tract Infection (Infections and infestations) | 9 | 9
Irritability (General disorders) | 6 | 11
Feeling Jittery (General disorders) | 2 | 11
Insomnia (Psychiatric disorders) | 4 | 12
Initial Insomnia (Psychiatric disorders) | 3 | 17
Anxiety (Psychiatric disorders) | 2 | 12
Decreased Appetite (Metabolism and nutrition disorders) | 7 | 25
Palpitations (Cardiac disorders) | 0 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI has the right to publish results of research and background information provided by SPONSOR necessary to include in publication of research results or for others to verify results. PI shall include a statement that creation of data was supported by SPONSOR. Prior to submission for publication/presentation, the INSTITUTION shall provide SPONSOR at least sixty (60) days for review.